CLINICAL TRIAL: NCT01704690
Title: Combination Treatment of S-1 With Paclitaxel Versus Paclitaxel+Cisplatin and 5-Fu+Cisplatin as First-line Treatment in Advanced Esophageal Cancer
Brief Title: Combination Treatment of S-1 With Paclitaxel in Advanced Esophageal Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The enrollment of the study is much slower than expected.
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhang, Head of Medical Oncology VIP-II department, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC001
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Chemotherapy; Efficacy; Toxicity
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); Paclitaxel; tegafur-gimeracil-oteracil; TP protocol; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- S-1 and Paclitaxel (Experimental): Patients in these arm will receive combination treatment of S-1 and paclitaxel. S-1, 80-120mg po, bid, from day 1 to day 14 Paclitaxel, 175mg/m2, IV infusion on day 1 Repeated every 21 days
  Interventions: Drug: S-1 and Paclitaxel
- Paclitaxel and Cisplatin (Active Comparator): Patients in these arm will receive combination treatment of paclitaxel and cisplatin.
  Paclitaxel, 175mg/m2, IV infusion on day 1 Cisplatin, 30 mg/m2, IV infusion on day 1 and day 2 Repeated every 21 days
  Interventions: Drug: Paclitaxel and Cisplatin
- 5-FU and Cisplatin (Active Comparator): Patients in these arm will receive combination treatment of 5-FU and cisplatin. 5-FU, 2500mg/m2, continue iv infusion for 120 hours Cisplatin, 35 mg/m2, IV infusion on day 1 and day 2 Repeated every 21 days
  Interventions: Drug: 5-FU and Cisplatin

INTERVENTIONS:
Drug: S-1 and Paclitaxel — S-1 and Paclitaxel are used in the S-1 and Paclitaxel arm.
  Other Names: TEYSUNO; TAXOL
  Arms: S-1 and Paclitaxel
Drug: Paclitaxel and Cisplatin — The paclitaxel and cisplatin combination will be used in the Paclitaxel and Cisplatin arm.
  Other Names: TAXOL; PLATINOL
  Arms: Paclitaxel and Cisplatin
Drug: 5-FU and Cisplatin — The cisplatin and 5-fluorouracil combination will be used in the Cisplatin and 5-FU arm.
  Other Names: 5-fluorouracil; PLATINOL
  Arms: 5-FU and Cisplatin

SUMMARY:
Esophageal cancer is one of the common malignant disease, especially in China. The annual incidence of esophageal squamous cell carcinoma is 260,000 with the motility of 210,000. The prognosis of esophageal cancer is very poor. About 50% of patients have advanced disease at diagnosis and the natural course is only 6-8 months with a 5-year survival rate of 5-7%. Though some patients received surgical treatment, disease will recurrent and metastasis in nearly 90% of the patients.

In past decades, there isn't much improvement of the outcome and survival of advanced esophageal cancer due to the lack of effective chemotherapy agents. The traditional chemotherapy drugs include 5-fluorouracil and cisplatin and the combination of them results in a 25-35% response rate in both first-line and palliative treatment. Paclitaxel plus cisplatin regiment is another promising treatment of esophageal cancer and have been proved effective in many studies. One of our previous study showed paclitaxel and cisplatin treatment resulted in encouraging response rate with manageable side-effects in 131 patients of advanced esophageal cancer.

However, the toxicities of paclitaxel and cisplatin limit their combination in clinic. For example, the polyoxyethylene castor oil paclitaxel could induce acute hypersensitivity reactions and neurotoxicity. Cisplatin could result in dysfunction of kidney and neurotoxicity. In addition, most of esophageal cancer patients are age 65 to 70. Many of them have simultaneously other diseases such as hypertension, diabetes, and chronic kidney disease which cause varying damages of renal function and limit the use of cisplatin in these patients. Therefore, it is urgent for doctors to seek an alternative of cisplatin in the combination chemotherapy treatment.

Therefore, the investigators designed this randomized clinical trial in which a novel combination of S-1 with paclitaxel is used to treat advanced esophageal cancer patients in compare with paclitaxel/cisplatin and 5-FU/cisplatin treatment to explore its efficacy and toxicity. The investigators hope this study will provide some clues for the treatment of esophageal cancer patients.

DETAILED DESCRIPTION:
Esophageal cancer is one of the common malignant tumors, especially in China and the annual incidence of esophageal squamous cell carcinoma is 260,000 with the motility of 210,000. In western countries, the incidence of esophageal adenocarcinoma (esophageal - gastric junction carcinoma) now dramatically increased than in the past. The pathological types of highest incidences are changing from esophageal squamous cell carcinoma (Esophageal Squamous Cell Carcinoma, ESCC) to esophageal adenocarcinoma (Esophageal adenocarcinoma, EAC) whose incidence is about 60-70%. But in Asia, esophageal squamous cell carcinoma is still the dominant pathological type, accounting for more than 95%. The prognosis of esophageal cancer is very poor. About 50% of patients have advanced disease at diagnosis and the natural course is only 6-8 months with a 5-year survival rate of 5-7%. In addition, though some patients received surgical treatment, disease will recurrent and metastasis in nearly 90% of the patients. For those patients in early stage (T1), there are still nearly 50% of patients relapse within 5 years. Therefore, in recent years, doctors and researchers in different countries are continued to seek effective treatment to improve the quality of life of patients with esophageal cancer and prolong survival.

In past decades, there isn't much improvement of the outcome and survival of advanced esophageal cancer due to the lack of effective chemotherapy agents. The traditional chemotherapy drugs to treat esophageal cancer include 5 - fluorouracil and cisplatin and the combination of them results in a 25-35% response rate in both first-line and palliative treatment. And this combing is still the traditional chemotherapy regimens and wildly used in clinical studies to treat both esophageal gland, squamous cell carcinoma of the clinical study.

Paclitaxel plus cisplatin regiment is another promising treatment of esophageal cancer and have been proved effective in a lot of studies. This combination has become a standard treatment of esophageal cancer, especially the esophageal squamous cell carcinoma. In one of our previous study, paclitaxel and cisplatin treatment showed encouraging clinical results with manageable side-effects in 131 patients of advanced esophageal cancer. These investigations have fully proved the efficacy and feasibility of the combination of paclitaxel with cisplatin regiment in the treatment of esophageal cancer. However, the lower solubility of paclitaxel limited its direct intravenous use. To solve this problem, the paclitaxel must inject with an addition of the surfactant polyoxyethylene castor oil. Polyoxyethylene castor oil paclitaxel could induce high incidence of acute hypersensitivity reactions, ie. severe allergic reactions, kidney damage, and neurotoxicity and cardiovascular toxicity which is characterized by axonal degeneration and demyelination. Though proper preventive treatment will greatly reduce the incidence of allergy, there are still a small number of patients have allergy reaction.

As the investigators all know, the main adverse of cisplatin is the renal toxicity. The peak age of esophageal cancer patients are age 65 to 70 and many of them have simultaneously other diseases such as hypertension, diabetes, and chronic kidney disease which cause varying damages of renal function and limit the use of cisplatin in these patients. Therefore, it is urgent and crucial for doctors to seek an alternative of cisplatin in the combination chemotherapy treatment. There haven't well designed large scale clinical trials to evidence the non-platinum treatment in esophageal cancer. Therefore, the investigators designed this randomized clinical trial in which a novel combination of S-1 with paclitaxel is used to treat advanced esophageal cancer patients in compare with paclitaxel/cisplatin and 5-FU/cisplatin treatment to explore its efficacy and toxicity. The investigators hope this study will provide some clues for the treatment of esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have histologically confirmed diagnosis of esophageal cancer without prior palliative treatment or an interval of at least 6 months from the last operation, adjuvant radiation therapy and adjuvant chemotherapy. If patients received adjuvant chemotherapy, paclitaxel and cisplatin must be excluded from the regiment or the total dosage of cisplatin must be less than 300mg/m2.
* - Patients must be 18 to 75 years old and both genders are eligible.
* - Patients must have measurable or evaluable disease with at least one tumor mass maximum diameter ≥10mm by multi-slice spiral CT or MR scan. If ordinary CT scan is used the tumor mass maximum diameter must ≥ 2cm. Imaging exam must be performed within 15 days from enrollment.
* - Patients must have an expected life expectancy of ≥ 3 months
* - Patients must have a performance status of ≥ 80 on the Karnofsky scale
* - Patients must have normal marrow function and the blood tests must be collected within 7 days from enrollment with a hemoglobin (HGB) of ≥90g/L, an white blood cell (WBC) counts of ≥4.0×109/L，a neutrophil count of ≥2.0×109/L, , a platelet count of ≥100×109/L, a total bilirubin (TBil) of ≤1.0 upper normal limitation (UNL), a creatinine (Cr) of ≤ 1.0 UNL, alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL, Alkaline phosphatase (AKP) ≤5.0 UNL. For patients with liver metastasis, the ASAT/ALAT must be ≤5.0 UNL.
* - Patients must have normal electrocardiogram results and no history of congestive heart failure.
* - Patients must be with good compliance and agree to accept follow-up of disease progression and adverse events.
* - Patients must give written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors

Exclusion Criteria:

* Patients who have received prior palliative treatment or less than 6 months from the last operation, adjuvant radiotherapy, adjuvant chemotherapy.
* Previous treatment regiment involve paclitaxel and S-1
* Tumor mass >10mm by CT or MR scan. The total area of metastatic tumor lesions in liver is over 50% of whole liver or the total area of metastatic tumor lesions in lung is over 25% of whole lung.
* Patients without measurable or evaluable disease, for example cavity effusion or diffusive metastasis of organs.
* Patients with history of other tumors except for those of cervical carcinoma in situ or skin basal cell carcinoma who had been completely treated and without relapse in last 5 years.
* Patients with serious diseases such as congestive heart failure, uncontrolled myocardial infarction and arrhythmia, liver failure and renal failure.
* Patients with only brain metastasis or bone metastasis
* Patients with chronic diarrhea
* Patients with neurological or psychiatric abnormalities including metastasis of the central nervous system that affect cognitive.
* Pregnant or lactated women (premenopausal women must give urine pregnancy test before enrollment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Every 2 cycles of treatment (average 6 weeks) up to 6cycles (assessed 18 weeks)
  The disease control rate (DCR) will be evaluated every 2 cycles (average 6 weeks) of treatment according to the RECIST 1.0 criteria until disease progression or finishing all 6 cycles of treatment.

SECONDARY OUTCOMES:
The median overall survival time | From date of randomization until the date of death from any cause (assessed up to 36 months)
  All the participants will receive chemotherapy very 3 weeks until disease progression. And after all 6 cycles of treatment, patients will be followed every 3 months until death from any cause or lost to follow up (up to 36 months). The median overall survival time will be measured using SPSS software version 17.0.
Median progression-free time | From date of randomization until the date of first documented progression or death from any cause (assessed up tp 36 months)
  All the participants will receive chemotherapy very 3 weeks until disease progression and the response will be evaluated every 2 cycles (about 6 weeks). And after all 6 cycles of treatment, patients will be followed and re-evaluated every 3 months until disease progression or death from any cause (up to 36 months). The median progression-free survival time will be measured using SPSS software version 17.0.
Number of Participants with Adverse Events and the degree of each adverse event | Participants will be followed every week during treatment and every 3 months during follow-up time (assessed up to 1 year)
  Both the number of subjects with adverse events and the degree of the adverse events of each participant according to NCI CTCAE version 3.0 will be recorded. And the outcome of each adverse event will be followed. The rate of adverse events will be compared in different arms.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhang, MD, Principal Investigator — Beijing Cancer Hospital, Peking University Cancer Hospital
Locations (1):
- Beijing Cancer Hospital, Peking University Cancer Hospital, Beijing, China

REFERENCES:
- [Background] Devesa SS, Blot WJ, Fraumeni JF Jr. Changing patterns in the incidence of esophageal and gastric carcinoma in the United States. Cancer. 1998 Nov 15;83(10):2049-53. PMID 9827707
- [Background] Bollschweiler E, Wolfgarten E, Gutschow C, Holscher AH. Demographic variations in the rising incidence of esophageal adenocarcinoma in white males. Cancer. 2001 Aug 1;92(3):549-55. doi: 10.1002/1097-0142(20010801)92:33.0.co;2-l. PMID 11505399
- [Background] Ilson DH. Oesophageal cancer: new developments in systemic therapy. Cancer Treat Rev. 2003 Dec;29(6):525-32. doi: 10.1016/s0305-7372(03)00104-x. PMID 14585262
- [Background] Anderson SE, Minsky BD, Bains M, Kelsen DP, Ilson DH. Combined modality therapy in esophageal cancer: the Memorial experience. Semin Surg Oncol. 2003;21(4):228-32. doi: 10.1002/ssu.10041. PMID 14648780
- [Background] Scheithauer W. Esophageal cancer: chemotherapy as palliative therapy. Ann Oncol. 2004;15 Suppl 4:iv97-100. doi: 10.1093/annonc/mdh911. No abstract available. PMID 15477344
- [Background] Koshy M, Esiashvilli N, Landry JC, Thomas CR Jr, Matthews RH. Multiple management modalities in esophageal cancer: combined modality management approaches. Oncologist. 2004;9(2):147-59. doi: 10.1634/theoncologist.9-2-147. PMID 15047919
- [Background] Westerterp M, Koppert LB, Buskens CJ, Tilanus HW, ten Kate FJ, Bergman JJ, Siersema PD, van Dekken H, van Lanschot JJ. Outcome of surgical treatment for early adenocarcinoma of the esophagus or gastro-esophageal junction. Virchows Arch. 2005 May;446(5):497-504. doi: 10.1007/s00428-005-1243-1. Epub 2005 Apr 19. PMID 15838647
- [Background] Enzinger PC, Ilson DH, Kelsen DP. Chemotherapy in esophageal cancer. Semin Oncol. 1999 Oct;26(5 Suppl 15):12-20. PMID 10566606
- [Background] Bleiberg H, Conroy T, Paillot B, Lacave AJ, Blijham G, Jacob JH, Bedenne L, Namer M, De Besi P, Gay F, Collette L, Sahmoud T. Randomised phase II study of cisplatin and 5-fluorouracil (5-FU) versus cisplatin alone in advanced squamous cell oesophageal cancer. Eur J Cancer. 1997 Jul;33(8):1216-20. doi: 10.1016/s0959-8049(97)00088-9. PMID 9301445
- [Background] Ilson DH, Forastiere A, Arquette M, Costa F, Heelan R, Huang Y, Kelsen DP. A phase II trial of paclitaxel and cisplatin in patients with advanced carcinoma of the esophagus. Cancer J. 2000 Sep-Oct;6(5):316-23. PMID 11079171
- [Background] Polee MB, Tilanus HW, Eskens FA, Hoekstra R, Van der Burg ME, Siersema PD, Stoter G, Van der Gaast A. Phase II study of neo-adjuvant chemotherapy with paclitaxel and cisplatin given every 2 weeks for patients with a resectable squamous cell carcinoma of the esophagus. Ann Oncol. 2003 Aug;14(8):1253-7. doi: 10.1093/annonc/mdg328. PMID 12881388
- [Background] Mu L, Feng SS. A novel controlled release formulation for the anticancer drug paclitaxel (Taxol): PLGA nanoparticles containing vitamin E TPGS. J Control Release. 2003 Jan 9;86(1):33-48. doi: 10.1016/s0168-3659(02)00320-6. PMID 12490371
- [Background] Mu L, Feng SS. Vitamin E TPGS used as emulsifier in the solvent evaporation/extraction technique for fabrication of polymeric nanospheres for controlled release of paclitaxel (Taxol). J Control Release. 2002 Apr 23;80(1-3):129-44. doi: 10.1016/s0168-3659(02)00025-1. PMID 11943393
- [Background] Lundberg BB, Risovic V, Ramaswamy M, Wasan KM. A lipophilic paclitaxel derivative incorporated in a lipid emulsion for parenteral administration. J Control Release. 2003 Jan 9;86(1):93-100. doi: 10.1016/s0168-3659(02)00323-1. PMID 12490375